CLINICAL TRIAL: NCT05347316
Title: Colchicine Effect on Perivascular Inflammation Index on Coronary CTA(COPIX Trial)
Brief Title: Colchicine Effect on Perivascular Inflammation Index on Coronary CTA
Acronym: COPIX
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Jr, MD PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC 5327/21/102
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerosis; Inflammatory Response; Coronary Disease
Keywords: Perivascular adipose tissue attenuation; Fat attenuation index; Colchicine; Coronary disease; Inflammation
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): 0.5 mg of colchicine daily for 12 months
  Interventions: Drug: Colchicine
- Placebo (No Intervention): Follow-up for 12 months

INTERVENTIONS:
Drug: Colchicine — 0.5 mg per day colchicine for 12 months
  Arms: Colchicine

SUMMARY:
Inflammation is an important pillar of atherogenesis in coronary disease. Studies have documented the prognostic power of measuring coronary perivascular adipose tissue attenuation (PVAT) and its good correlation as an early inflammatory biomarker in the atherogenesis process, in addition to being a predictor for cardiovascular events in the future. Colchicine, a medication with well-documented anti-inflammatory action and with an impact on reducing cardiovascular outcomes, may have an action in reducing FAI (fat attenuation index). This study aims to evaluate the effect of colchicine in reducing coronary perivascular inflammation.

DETAILED DESCRIPTION:
A single-center, prospective, single-blind randomized study to evaluate the efficacy of colchicine versus placebo in patients with documented FAI ≥ -70.1 HU of the proximal segment of the right coronary artery and/ou left anterior descending coronary artery and non-calcified or mixed plaques on coronary angiography performed electively after 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes over 18 years of age;
* Patients undergoing coronary CT angiography from May/2021
* CT angiography showing non-calcified or mixed coronary plaques and high FAI value (> -70.1 HU) in the proximal segment of the right and/or anterior descending coronary artery with
* Willing and able (in the opinion of the investigators) to fulfill all study requirements

Exclusion Criteria:

* Past history of acute myocardial infarction
* History of percutaneous or surgical myocardial revascularization
* History of previous cardiac surgery or congenital heart disease
* Current use of colchicine
* Autoimmune disease requiring immunosuppressive therapy or current use of systemic corticosteroid therapy
* Active neoplasm with indication of surgery, chemotherapy or radiation in the last 12 months (patients with a history of neoplasm and who underwent curative surgery without need for treatment in the last 12 months will be allowed)
* Inflammatory bowel disease or chronic diarrhea
* Clinically significant non-transient hematologic abnormalities
* Renal dysfunction (GFR < 30 mL/min/1.73 m² and/or serum creatinine > 2.5 mg/dL or < 220 µmol/l)
* Severe liver disease (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3x ULN in the last 6 months)
* Drug addiction or alcoholism
* History of clinically significant sensitivity to colchicine
* Inability to sign the informed consent form
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — over 18 years
Enrollment: 40 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of FAI in both groups after 12-month follow-up | 12 months

SECONDARY OUTCOMES:
Evaluation of the variation total atheroma volume | 12 months
Evaluation of low attenuation plate volume variation; | 12 months
Occurrence of general death | 12 months
Occurrence of cardiovascular death | 12 months
Occurrence of acute myocardial infarction | 12 months
Occurrence of stroke | 12 months
Occurrence of need for myocardial revascularization | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute - University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No